CLINICAL TRIAL: NCT06395987
Title: Result Of Use Of Wide Awake Local Anaesthesia In Fixation Of Ankle Fractures
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Sayed Shahata, Assistant Lecturer, Assiut University
Other Study IDs: WALANT FOR ANKLE FRACTURES
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Local Anesthesia
Keywords: Wide_awake

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Wide Awake Local Anaesthesia In Fixation Of Ankle Fractures. — Use Of Wide Awake Local Anaesthesia In Fixation Of Ankle Fractures.

SUMMARY:
to assess the success of wide-awake local anaesthesia In fixation of ankle fractures

DETAILED DESCRIPTION:
The wide-awake local anesthesia with no tourniquet provides an alternative method for the existing anesthesia methods including general anesthesia, intrathecal, epidural anesthesia, peripheral nerve block and local anesthesia with intravenous sedation. Each method of them has its inherent risks and costs.

The wide-awake local anesthesia has few risks for the patient and can be used in satisfaction where other types of anesthesia particularly general anesthesia are contraindicated.

This method is safe, effective and provides satisfactory pain and anxiety scores. Patients don't have to stay for a long time after surgery. It allows the surgery to be done without tourniquet due to the use of epinephrine and this avoids the complication of tourniquet and allows the surgery to be done safely in cases of limb vascular insufficiency and in diabetic patients where tourniquet usage is not favorable.

Wide awake local anesthesia method for ankle fracture management is not a novel idea; it was previously investigated in one study but the limitation of this study that it was retrospective study with small sample size and without control group treated with other anesthetic modalities.

There is concern that the use of lidocaine in hematoma block is harmful for joint cartilage. Excess use of epinephrine may cause excessive vasoconstriction and cyanosis of fingers . Neuropathic complication are notably high during the early postsurgical period .

Wide-awake anesthesia is delivered by the surgeon . The role of anesthetic team, if needed, is monitoring the vital signs and in case of failure of wide-awake and prolonged time of surgery .

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with unstable ankle fracture who need fixation presenting to the Trauma Unit of Assiut University Hospital with the following criteria:

  1. Age ≥ 18 years.
  2. Isolated ankle fracture in one or both lower limbs.

Exclusion Criteria:

1. patients< 18 years.
2. Patients with uncontrolled diabetes mellitus.
3. open fractures.
4. Associated fractures in the lower limbs(Spinal anaesthesia will be more suitable in multiple fractures)
5. Fractures managed by closed contact casting.
6. Patients with dementia and psychological disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to assess the success of wide-awake local anaesthesia In fixation of ankle fractures.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-05-16 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
• Success of wide-awake local anaesthesia in fixation of ankle fractures by measuring the amount of failure of wide awake local anesthesia | Follow up for 6 months to assess if there is any complications .
  Measure the success rate of wide awake inrelarion to failed cases

CONTACTS AND LOCATIONS:
Overall Officials: Wael Youssef El-Adly, Professor, Study Chair — Assiut University

REFERENCES:
- [Background] Hansen E, Eshelman MR, Cracchiolo A 3rd. Popliteal fossa neural blockade as the sole anesthetic technique for outpatient foot and ankle surgery. Foot Ankle Int. 2000 Jan;21(1):38-44. doi: 10.1177/107110070002100107. PMID 10710260
- [Background] Lalonde D, Martin A. Tumescent local anesthesia for hand surgery: improved results, cost effectiveness, and wide-awake patient satisfaction. Arch Plast Surg. 2014 Jul;41(4):312-6. doi: 10.5999/aps.2014.41.4.312. Epub 2014 Jul 15. PMID 25075350
- [Background] Wright J, MacNeill AL, Mayich DJ. A prospective comparison of wide-awake local anesthesia and general anesthesia for forefoot surgery. Foot Ankle Surg. 2019 Apr;25(2):211-214. doi: 10.1016/j.fas.2017.10.015. Epub 2017 Nov 6. PMID 29409279
- [Background] Thomson CJ, Lalonde DH, Denkler KA, Feicht AJ. A critical look at the evidence for and against elective epinephrine use in the finger. Plast Reconstr Surg. 2007 Jan;119(1):260-266. doi: 10.1097/01.prs.0000237039.71227.11. PMID 17255681
- [Background] Anderson JG, Bohay DR, Maskill JD, Gadkari KP, Hearty TM, Braaksma W, Padley MA, Weaver KT. Complications After Popliteal Block for Foot and Ankle Surgery. Foot Ankle Int. 2015 Oct;36(10):1138-43. doi: 10.1177/1071100715589741. Epub 2015 Jun 24. PMID 26109605
- [Background] Lalonde D. Minimally invasive anesthesia in wide awake hand surgery. Hand Clin. 2014 Feb;30(1):1-6. doi: 10.1016/j.hcl.2013.08.015. Epub 2013 Nov 9. PMID 24286736
- [Background] Pires Neto PJ, Moreira LA, Las Casas PP. Is it safe to use local anesthesia with adrenaline in hand surgery? WALANT technique. Rev Bras Ortop. 2017 Jul 19;52(4):383-389. doi: 10.1016/j.rboe.2017.05.006. eCollection 2017 Jun-Jul. PMID 28884094
- [Background] Lalonde DH, Wong A. Dosage of local anesthesia in wide awake hand surgery. J Hand Surg Am. 2013 Oct;38(10):2025-8. doi: 10.1016/j.jhsa.2013.07.017. Epub 2013 Sep 8. No abstract available. PMID 24021739